CLINICAL TRIAL: NCT04655612
Title: Seroprevalence Study of CoV-2-SARS (COVID-19) Infection in Patients With Chronic Inflammatory Rheumatic Diseases
Acronym: COVID-RIC1
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0624
Record Dates: First submitted 2020-12-03; First posted 2020-12-07 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; SARS-CoV Infection; Rheumatoid Arthritis; Spondyloarthritis; Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: COVID-19; SARS-COV-2 infection; Rheumatoid arthritis; Spondyloarthritis
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Arthritis, Rheumatoid; Spondylarthritis; Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of SARS-CoV-2 infection in chronic inflammatory rheumatic diseases has not yet been widely reported, and has been evaluated only in symptomatic patient samples. The proportion of asymptomatic or mildly symptomatic patients is unknown, in patients who share common symptoms with CoV-2-SARS infection. Our objective is to describe the prevalence of seroconversion to CoV-2-SARS by consecutive screening in routine care of patients with chronic inflammatory rheumatism with serological testing

DETAILED DESCRIPTION:
The prevalence of SARS-CoV-2 infection in chronic inflammatory rheumatic diseases has not yet been widely reported, and has been evaluated only in symptomatic patient samples. The proportion of asymptomatic or mildly symptomatic patients is unknown, in patients who share common symptoms with CoV-2-SARS infection.

Some treatments for chronic inflammatory rheumatisms such as TNF inibitors appear to have a protective effect against severe forms of COVID-19, while corticosteroids or other immunosuppressants may be associated with a higher prevalence of severe forms of COVID-19.

Our objective is to describe the prevalence of seroconversion to CoV-2-SARS by consecutive screening in routine care of out and inpatients with chronic inflammatory rheumatism (i.e. rheumatoid arthritis, axial spondyloarthritis and psoriatic arthritis) by serological testing and to compare prevalence according to type of chronic inflammatory rheumatism, DMARD class and symptomatic treatment (corticosteroid therapy, NSAIDs).

ELIGIBILITY:
Inclusion criteria:

- Patient with chronic inflammatory rheumatic disease (i.e. rheumatoid arthritis, psoriatic rheumatism, axial spondyloarthritis), Coming for consultation or hospitalization as part of the usual follow-up of his condition

Exclusion criteria:

- Adult patient under legal protection (guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive outpatients and inpatients with inflammatory chronic rheumatism disease
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with inflammatory chronic rheumatic diseases with positive SARS-CoV-2 serodiagnosis | 1 day
  Proportion of patients with inflammatory chronic rheumatic diseases with positive SARS-CoV-2 serodiagnosis

SECONDARY OUTCOMES:
Proportion of patients with a positive CoV-2 SARS serodiagnosis according to current treatments. | 1 day
  Proportion of patients with a positive CoV-2 SARS serodiagnosis according to current treatments.
Proportion of patients with a positive CoV-2 SARS serodiagnosis according to type of chronic inflammatory rheumatic disease | 1 day
  Proportion of patients with a positive CoV-2 SARS serodiagnosis according to type of chronic inflammatory rheumatic disease
Proportion of patients with a positive CoV-2 SARS serodiagnosis according to demographic characteristics | 1 day
  Proportion of patients with a positive CoV-2 SARS serodiagnosis according to demographic characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Morel, MD, PhD, Study Director — UH MONTPELLIER; Thao Pham, MD, PhD, Principal Investigator — AP-HM
Locations (1):
- Centre hopsitalier universitaire de Montpellier, Montpellier, Occitanie, France

IPD SHARING:
Plan to Share IPD: Undecided
NC